CLINICAL TRIAL: NCT01710358
Title: A Randomized, Double-Blind, Placebo- and Active-Controlled, Phase 3 Study Evaluating the Efficacy and Safety of Baricitinib in Patients With Moderately to Severely Active Rheumatoid Arthritis Who Have Had an Inadequate Response to Methotrexate Therapy
Brief Title: A Study in Moderate to Severe Rheumatoid Arthritis
Acronym: RA-BEAM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13978; I4V-MC-JADV (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-10-17; First posted 2012-10-19 (Estimated); Results first posted 2017-08-15 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab; baricitinib; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Placebo administered orally once daily through Week 24 and placebo administered by subcutaneous (SC) injection every 2 weeks through Week 50.
  At Week 24, participants were given baricitinib 4 milligram (mg) orally once daily through Week 52.
  Starting at Week 16, participants who were nonresponders were rescued with baricitinib 4 mg orally daily through Week 52.
  Participants continued to take background methotrexate (MTX) therapy throughout study.
  Interventions: Drug: Methotrexate; Drug: Adalimumab Placebo; Drug: Baricitinib Placebo
- Baricitinib (Experimental): Baricitinib 4 mg administered orally once daily through Week 52 and an adalimumab placebo SC injection every 2 weeks through Week 50.
  Starting at Week 16, nonresponder participants originally randomized to baricitinib continued to receive baricitinib 4 mg administered orally once daily through Week 52.
  Participants continued to take background methotrexate (MTX) therapy throughout study.
  Interventions: Drug: Baricitinib; Drug: Methotrexate; Drug: Adalimumab Placebo
- Adalimumab (Active Comparator): Adalimumab 40 mg administered by SC injection every 2 weeks through Week 50 and baricitinib placebo orally once daily through Week 52.
  Starting at Week 16, participants who were nonresponders were rescued with baricitinib 4 mg orally once daily through Week 52.
  Participants continued to take background methotrexate (MTX) therapy throughout study.
  Interventions: Drug: Adalimumab; Drug: Methotrexate; Drug: Baricitinib Placebo

INTERVENTIONS:
Drug: Adalimumab — Administered SC
  Arms: Adalimumab
Drug: Baricitinib — Administered orally
  Other Names: LY 3009104
  Arms: Baricitinib
Drug: Methotrexate — Administered orally
Drug: Adalimumab Placebo — Adalimumab placebo administered SC.
  Arms: Baricitinib; Placebo
Drug: Baricitinib Placebo — Baricitinib placebo administered orally.
  Arms: Adalimumab; Placebo

SUMMARY:
The purpose of this study is to determine whether baricitinib is superior to placebo in the treatment of participants with moderately to severely active Rheumatoid Arthritis (RA) who have had an inadequate response to methotrexate (MTX) treatment.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of adult-onset Rheumatoid Arthritis (RA) as defined by the American College of Rheumatology/ European League Against Rheumatism (ACR/EULAR) 2010 Criteria for the Classification of RA
* Have moderately to severely active RA defined as the presence of at least 6/68 tender joints and at least 6/66 swollen joints
* Have a C-reactive protein (CRP) or high-sensitivity C-reactive protein (hsCRP) measurement ≥6 milligram per Liter (mg/L)
* Have had regular use of methotrexate (MTX) for at least the 12 weeks prior to study entry at a dose that is considered acceptable to adequately assess clinical response.
* Have at least 1 joint erosion in hand, wrist, or foot joints based on radiographic interpretation by the central reader and be rheumatoid factor or anticyclic citrullinated peptide (anti-CCP) antibody positive; or have at least 3 joint erosions in hand, wrist, or foot joints based on radiographic interpretation by the central reader regardless of rheumatoid factor or anti-CCP antibody status

Exclusion Criteria:

* Are currently receiving corticosteroids at doses >10 mg of prednisone per day (or equivalent) or have been receiving an unstable dosing regimen of corticosteroids within 2 weeks of study entry or within 6 weeks of planned randomization
* Have started treatment with non-steroidal anti-inflammatory drugs (NSAIDs) or have been receiving an unstable dosing regimen of NSAIDs within 2 weeks of study entry or within 6 weeks of planned randomization
* Are currently receiving concomitant treatment with MTX, hydroxychloroquine, and sulfasalazine or combination of any 3 conventional disease-modifying antirheumatic drugs (cDMARDs)
* Are currently receiving or have received cDMARDs (eg, gold salts, cyclosporine, azathioprine, or any other immunosuppressives) other than MTX, hydroxychloroquine (up to 400 mg/day), or sulfasalazine (up to 3000 mg/day) within 4 weeks prior to study entry
* Have received leflunomide in the 12 weeks prior to study entry
* Have started a new physiotherapy treatment for RA in the 2 weeks prior to study entry
* Have ever received any biologic disease-modifying antirheumatic drugs (DMARD)
* Have received interferon therapy within 4 weeks prior to study entry or are anticipated to require interferon therapy during the study
* Have received any parenteral corticosteroid administered by intramuscular or intravenous injection within 2 weeks prior to study entry or within 6 weeks prior to planned randomization or are anticipated to require parenteral injection of corticosteroids during the study
* Have had 3 or more joints injected with intraarticular corticosteroids or hyaluronic acid within 2 weeks prior to study entry or within 6 weeks prior to planned randomization
* Have any condition or contraindication for adalimumab that would preclude the participant from participating in this protocol
* Have active fibromyalgia that would make it difficult to appropriately assess RA activity for the purposes of this study
* Have a diagnosis of any systemic inflammatory condition other than RA such as, but not limited to, juvenile chronic arthritis, spondyloarthropathy, Crohn's disease, ulcerative colitis, psoriatic arthritis, active vasculitis or gout(participants with secondary Sjögren's syndrome are not excluded)
* Have a diagnosis of Felty's syndrome
* Have had any major surgery within 8 weeks prior to study entry or will require major surgery during the study that, in the opinion of the investigator in consultation with Lilly or its designee, would pose an unacceptable risk to the participant
* Have experienced any of the following within 12 weeks of study entry: myocardial infarction, unstable ischemic heart disease, stroke, or New York Heart Association Stage IV heart failure
* Have a history or presence of cardiovascular, respiratory, hepatic, gastrointestinal, endocrine, hematological, neurological, or neuropsychiatric disorders or any other serious and/or unstable illness that, in the opinion of the investigator, could constitute a risk when taking investigational product or could interfere with the interpretation of data
* Are largely or wholly incapacitated permitting little or no self-care, such as being bedridden or confined to a wheelchair
* have a history of, lymphoproliferative disease; or have signs or symptoms suggestive of possible lymphoproliferative disease, including lymphadenopathy or splenomegaly; or have active primary or recurrent malignant disease; or have been in remission from clinically significant malignancy for <5 years
* Have been exposed to a live vaccine within 12 weeks prior to planned randomization or are expected to need/receive a live vaccine during the course of the study (with the exception of herpes zoster vaccination)
* Have a current or recent clinically serious viral, bacterial, fungal, or parasitic infection
* Have had symptomatic herpes zoster infection within 12 weeks prior to study entry
* Have a history of disseminated/complicated herpes zoster (eg, multidermatomal involvement, ophthalmic zoster, central nervous system involvement, or postherpetic neuralgia)
* Are immunocompromised and, in the opinion of the investigator, are at an unacceptable risk for participating in the study
* Have a history of active hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV)
* Have screening laboratory test values, including thyroid-stimulating hormone (TSH), outside the reference range for the population or investigative site that, in the opinion of the investigator, pose an unacceptable risk for the participant's participation in the study
* Have screening electrocardiogram (ECG) abnormalities that, in the opinion of the investigator or the sponsor, are clinically significant and indicate an unacceptable risk for the participant's participation in the study
* Have symptomatic herpes simplex at the time of study enrollment
* Have evidence of active or latent tuberculosis (TB)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1307 (Actual)
Dates: Start 2012-10; Primary Completion 2015-03 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (211):
- United States (45):
  - Arizona Arthritis & Rheumatology Research, Glendale, Arizona
  - Sun Valley Arthritis Center, LTD, Peoria, Arizona
  - Valley Arthritis Care, LLC, Phoenix, Arizona
  - University of Boards Regent, Tucson, Arizona
  - Valley Endocrine, Fresno, Fresno, California
  - Desert Medical Advances, Palm Desert, California
  - Pacific Arthritis Center, Santa Maria, California
  - Inlande Rheumatology Clinical Trials, Upland, California
  - Boulder Medical Center, Boulder, Colorado
  - Clinical Research Center of CT/NY, Danbury, Connecticut
  - New England Research Associates, Trumbull, Connecticut
  - Delaware Arthritis, Lewes, Delaware
  - Orthopedic Research Institute, Boynton Beach, Florida
  - Jeffrey Alper, M.D., Naples, Florida
  - Sun Coast Clinical Research, Inc, New Port Richey, Florida
  - Rheumatology Associates of Central Florida, Orlando, Florida
  - Integral Rheumatology & Immunology Specialists, Plantation, Florida
  - McIlwain Medical Group, Tampa, Florida
  - Indiana University Health, Indianapolis, Indiana
  - Diagnostic Rheumatology and Research, Indianapolis, Indiana
  - Goldpoint Clinical Research LLC, Indianapolis, Indiana
  - West Michigan Rheumatology, Grand Rapids, Michigan
  - University of Missouri, Columbia, Missouri
  - Dr. George Timothy Kelly, Las Vegas, Nevada
  - (AOA) Arthritis & Osteoporosis Associates, Freehold, New Jersey
  - Bio Behavioral Health, Toms River, New Jersey
  - Drug Trials of America, Hartsdale, New York
  - Asheville Rheumatology & Osteoporosis Research Assoc, PA, Asheville, North Carolina
  - Paramount Medical Research, Middleburg Heights, Ohio
  - Health Research Institute, Oklahoma City, Oklahoma
  - Healthcare Research Consultant, Tulsa, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - East Penn Rheumatology, Bethlehem, Pennsylvania
  - Clinical Research Center of Reading, LLP, Wyomissing, Pennsylvania
  - Carolina Rheumatology and Neurology Associates, Myrtle Beach, South Carolina
  - Metroplex Clinical Research Center, Dallas, Texas
  - Pioneer Research Solutions, Houston, Texas
  - Accurate Clinical Research, Houston, Texas
  - Arthritis & Osteoporosis Associates LLP, Lubbock, Texas
  - Accurate Clinical Research, Nassau Bay, Texas
  - Accurate Clinical Research, Webster, Texas
  - Center for Arthritis and Rheumatic Diseases, PC, Chesapeake, Virginia
  - The Seattle Arthritis Clinic, Seattle, Washington
  - Vancouver Clinic, Vancouver, Washington
  - Rheumatology and Immunotherapy Center, Franklin, Wisconsin
- Argentina (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bahía Blanca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Caba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Córdoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mar del Plata
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Quilmes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rosario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Fernando
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Miguel de Tucumán
- Belgium (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brussels
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Genk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Merksem
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mons
- Canada (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kelowna, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Victoria, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kitchener, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Catherines, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toronto, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Trois-Rivières, Quebec
- China (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beijing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bengbu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Changsha
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guangzhou
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hefei
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jinan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shanghai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wuhan
- Croatia (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Varaždin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zagreb
- Czechia (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brno
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bruntál
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hustopeče
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ostrava
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ostrava - Trebovice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pardubice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prague
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Uherské Hradiště
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zlín
- France (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cahors
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Limoges
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montpellier
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nantes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orléans
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poitiers
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Strasbourg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Thionville
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tours
- Germany (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cologne
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gommern
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Herne
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Würzburg
- Greece (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Athens
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heraklion
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Larissa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marousi
- Hungary (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Budapest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kiskunhalas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nyíregyháza
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Székesfehérvár
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Veszprém
- Japan (28):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aichi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hiroshima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hokkaido
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyōgo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ibaraki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Japan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kagoshima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kumamoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mie
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagano
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagasaki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Niigata
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Numakunai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Okayama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Okinawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ōita
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saga
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saitama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shizuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tochigi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toyama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yamaguchi
- Latvia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Liepāja
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Riga
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valmiera
- Lithuania (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kaunas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Klaipėda
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Šiauliai
- Mexico (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guadalajara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexicali
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mérida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., México
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Luis Potosí City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tijuana
- Poland (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bydgoszcz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Elblag
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gdansk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Katowice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lodz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nadarzyn
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
- Portugal (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lisbon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Porto
- Puerto Rico (4):
  - Ramon L. Ortega Colon, Carolina
  - Office of Dr. Ramon Toro, San Germán
  - Mindful Medical Research, San Juan
  - Latin Clinical Trial Center, Santurce
- Romania (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cluj-Napoca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Constanța
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lasi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oradea
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Târgu Mureş
- Russia (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Korolyov
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ryazan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Petersburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saratov
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ulyanovsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yaroslavl
- Slovakia (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bratislava
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Partizánske
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spišská Nová Ves
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Topoľčany
- Slovenia (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ljubljana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Maribor
- South Africa (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Durban
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greenacres
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pinelands
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stellenbosch
- South Korea (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daegu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daejeon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gwangju
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Incheon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Suwon
- Spain (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bilbao
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., L'Hospitalet de Llobregat
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sabadell
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santander
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seville
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valencia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Villajoyosa
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fribourg, Switzerland
- Taiwan (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kaohsiung City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Neihu Taipei
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taichung
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yongkang District
- United Kingdom (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London, England
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London, Greater London
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Basingstoke, Hampshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Southampton, Hants
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aberdeen, Scotland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., North Shields, Tyneside
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bradford, West Yorkshire

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Landewe R, Sun L, Chen YF, Daojun M, van der Heijde D. Robust analyses for radiographic progression in rheumatoid arthritis. RMD Open. 2023 Apr;9(2):e002543. doi: 10.1136/rmdopen-2022-002543. PMID 37015757
- [Derived] Taylor PC, Takeuchi T, Burmester GR, Durez P, Smolen JS, Deberdt W, Issa M, Terres JR, Bello N, Winthrop KL. Safety of baricitinib for the treatment of rheumatoid arthritis over a median of 4.6 and up to 9.3 years of treatment: final results from long-term extension study and integrated database. Ann Rheum Dis. 2022 Mar;81(3):335-343. doi: 10.1136/annrheumdis-2021-221276. Epub 2021 Oct 27. PMID 34706874
- [Derived] van der Heijde D, Kartman CE, Xie L, Beattie S, Schlichting D, Mo D, Durez P, Tanaka Y, Fleischmann R. Radiographic Progression of Structural Joint Damage Over 5 Years of Baricitinib Treatment in Patients With Rheumatoid Arthritis: Results From RA-BEYOND. J Rheumatol. 2022 Feb;49(2):133-141. doi: 10.3899/jrheum.210346. Epub 2021 Sep 15. PMID 34526397
- [Derived] Emery P, Tanaka Y, Cardillo T, Schlichting D, Rooney T, Beattie S, Helt C, Smolen JS. Temporary interruption of baricitinib: characterization of interruptions and effect on clinical outcomes in patients with rheumatoid arthritis. Arthritis Res Ther. 2020 May 15;22(1):115. doi: 10.1186/s13075-020-02199-8. PMID 32414425
- [Derived] Schlueter M, Finn E, Diaz S, Dilla T, Inciarte-Mundo J, Fakhouri W. Cost-effectiveness analysis of baricitinib versus adalimumab for the treatment of moderate-to-severe rheumatoid arthritis in Spain. Clinicoecon Outcomes Res. 2019 Jun 6;11:395-403. doi: 10.2147/CEOR.S201621. eCollection 2019. PMID 31239736
- [Derived] Michaud K, Pope JE, Emery P, Zhu B, Gaich CL, DeLozier AM, Zhang X, Dickson CL, Smolen JS. Relative Impact of Pain and Fatigue on Work Productivity in Patients with Rheumatoid Arthritis from the RA-BEAM Baricitinib Trial. Rheumatol Ther. 2019 Sep;6(3):409-419. doi: 10.1007/s40744-019-0164-4. Epub 2019 Jun 21. PMID 31228100
- [Derived] Tanaka Y, Fautrel B, Keystone EC, Ortmann RA, Xie L, Zhu B, Issa M, Patel H, Gaich CL, de Bono S, Rooney TP, Taylor PC. Clinical outcomes in patients switched from adalimumab to baricitinib due to non-response and/or study design: phase III data in patients with rheumatoid arthritis. Ann Rheum Dis. 2019 Jul;78(7):890-898. doi: 10.1136/annrheumdis-2018-214529. Epub 2019 Apr 30. PMID 31040122
- [Derived] Bingham CO 3rd, Gaich CL, DeLozier AM, Engstrom KD, Naegeli AN, de Bono S, Banerjee P, Taylor PC. Use of daily electronic patient-reported outcome (PRO) diaries in randomized controlled trials for rheumatoid arthritis: rationale and implementation. Trials. 2019 Mar 22;20(1):182. doi: 10.1186/s13063-019-3272-0. PMID 30902094
- [Derived] Combe B, Balsa A, Sarzi-Puttini P, Tony HP, de la Torre I, Rogai V, Durand F, Witt S, Zhong J, Dougados M. Efficacy and safety data based on historical or pre-existing conditions at baseline for patients with active rheumatoid arthritis who were treated with baricitinib. Ann Rheum Dis. 2019 Aug;78(8):1135-1138. doi: 10.1136/annrheumdis-2018-214261. Epub 2019 Mar 6. No abstract available. PMID 30842122
- [Derived] Smolen JS, Genovese MC, Takeuchi T, Hyslop DL, Macias WL, Rooney T, Chen L, Dickson CL, Riddle Camp J, Cardillo TE, Ishii T, Winthrop KL. Safety Profile of Baricitinib in Patients with Active Rheumatoid Arthritis with over 2 Years Median Time in Treatment. J Rheumatol. 2019 Jan;46(1):7-18. doi: 10.3899/jrheum.171361. Epub 2018 Sep 15. PMID 30219772
- [Derived] Tanaka Y, McInnes IB, Taylor PC, Byers NL, Chen L, de Bono S, Issa M, Macias WL, Rogai V, Rooney TP, Schlichting DE, Zuckerman SH, Emery P. Characterization and Changes of Lymphocyte Subsets in Baricitinib-Treated Patients With Rheumatoid Arthritis: An Integrated Analysis. Arthritis Rheumatol. 2018 Dec;70(12):1923-1932. doi: 10.1002/art.40680. Epub 2018 Oct 22. PMID 30058112
- [Derived] Wells AF, Greenwald M, Bradley JD, Alam J, Arora V, Kartman CE. Baricitinib in Patients with Rheumatoid Arthritis and an Inadequate Response to Conventional Disease-Modifying Antirheumatic Drugs in United States and Rest of World: A Subset Analysis. Rheumatol Ther. 2018 Jun;5(1):43-55. doi: 10.1007/s40744-018-0110-x. Epub 2018 Apr 21. PMID 29680881
- [Derived] Taylor PC, Kremer JM, Emery P, Zuckerman SH, Ruotolo G, Zhong J, Chen L, Witt S, Saifan C, Kurzawa M, Otvos JD, Connelly MA, Macias WL, Schlichting DE, Rooney TP, de Bono S, McInnes IB. Lipid profile and effect of statin treatment in pooled phase II and phase III baricitinib studies. Ann Rheum Dis. 2018 Jul;77(7):988-995. doi: 10.1136/annrheumdis-2017-212461. Epub 2018 Feb 20. PMID 29463520
- [Derived] Keystone EC, Taylor PC, Tanaka Y, Gaich C, DeLozier AM, Dudek A, Zamora JV, Cobos JAC, Rooney T, Bono S, Arora V, Linetzky B, Weinblatt ME. Patient-reported outcomes from a phase 3 study of baricitinib versus placebo or adalimumab in rheumatoid arthritis: secondary analyses from the RA-BEAM study. Ann Rheum Dis. 2017 Nov;76(11):1853-1861. doi: 10.1136/annrheumdis-2017-211259. Epub 2017 Aug 10. PMID 28798049
- [Derived] Taylor PC, Keystone EC, van der Heijde D, Weinblatt ME, Del Carmen Morales L, Reyes Gonzaga J, Yakushin S, Ishii T, Emoto K, Beattie S, Arora V, Gaich C, Rooney T, Schlichting D, Macias WL, de Bono S, Tanaka Y. Baricitinib versus Placebo or Adalimumab in Rheumatoid Arthritis. N Engl J Med. 2017 Feb 16;376(7):652-662. doi: 10.1056/NEJMoa1608345. PMID 28199814

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who did not respond (nonresponders) to study drug were eligible for rescue treatment beginning at Week16. Participants not rescued at Week 16 may be rescued at the discretion of the investigator anytime thereafter.
  Nonresponders were defined as lack of improvement of at least 20% in both tender joint count and swollen joint count.
Groups:
- Placebo: Placebo administered orally (PO) once daily (QD) through Week 24 and placebo administered by subcutaneous (SC) injection every 2 weeks through Week 50.
  At Week 24, participants were given baricitinib 4 milligram (mg) orally once daily through Week 52.
  Starting at Week 16, participants who were nonresponders were rescued with baricitinib 4 mg orally once daily through Week 52.
  Participants continued to take background methotrexate (MTX) therapy throughout study.
- Baricitinib: Baricitinib 4 mg administered orally once daily through Week 52 and an adalimumab placebo SC injection every 2 weeks through Week 50.
  Starting at Week 16, nonresponder participants originally randomized to baricitinib continued to receive baricitinib 4 mg administered orally once daily through Week 52.
  Participants continued to take background MTX therapy throughout study.
- Adalimumab: Adalimumab 40 mg administered by SC injection every 2 weeks through Week 50 and baricitinib placebo orally once daily through Week 52.
  Starting at Week 16, participants who were nonresponders were rescued with baricitinib 4 mg orally once daily through Week 52.
  Participants continued to take background MTX therapy throughout study.
Period: Treatment Period Part A (Weeks 0 to 24)
Arm/Group | Placebo | Baricitinib | Adalimumab
Started | 489 | 488 | 330
Received at Least 1 Dose of Study Drug | 488 | 487 | 330
Rescued | 128 | 35 | 40
Completed | 438 (Includes all participants rescued during Part A.) | 459 (Includes all participants rescued during Part A.) | 307 (Includes all participants rescued during Part A.)
Not Completed | 51 | 29 | 23
Not completed — Adverse Event | 15 | 18 | 7
Not completed — Death | 0 | 2 | 0
Not completed — Entry Criteria Not Met | 0 | 1 | 1
Not completed — Lack of Efficacy | 15 | 1 | 3
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Sponsor Decision | 4 | 0 | 0
Not completed — Withdrawal by Subject | 15 | 5 | 12
Not completed — Randomized But Not Treated | 1 | 1 | 0
Period: Treatment Period Part B (Weeks 24 to 52)
Arm/Group | Placebo | Baricitinib | Adalimumab
Started | 310 (Excludes participants rescued during Part A.) | 424 (Excludes participants rescued during Part A.) | 267 (Excludes participants rescued during Part A.)
Received at Least 1 Dose of Study Drug | 306 (Participants originally randomized to placebo received baricitinib during Part B.) | 424 | 267
Rescued | 5 | 8 | 11
Completed | 294 (Includes all participants rescued during Part B.) | 402 (Includes all participants rescued during Part B.) | 252 (Includes all participants rescued during Part B.)
Not Completed | 16 | 22 | 15
Not completed — Adverse Event | 10 | 16 | 5
Not completed — Death | 1 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Sponsor Decision | 1 | 2 | 0
Not completed — Withdrawal by Subject | 4 | 3 | 7
Period: Rescue Period
Arm/Group | Placebo | Baricitinib | Adalimumab
Started | 0 (Participants who were nonresponders based on tender/swollen joint count entered into rescue group.) | 227 (Baricitinib 4 mg administered PO QD through Week 52. Participants continued background MTX therapy.) | 0 (Participants who were nonresponders based on tender/swollen joint count entered into rescue group.)
Completed | 0 | 196 | 0
Not Completed | 0 | 31 | 0
Not completed — Adverse Event | 0 | 15 | 0
Not completed — Death | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 7 | 0
Not completed — Withdrawal by Subject | 0 | 8 | 0
Period: Follow-up Period
Arm/Group | Placebo | Baricitinib | Adalimumab
Started | 33 (Participants from treatment who entered the post-treatment follow-up period.) | 76 (Rescued participants who entered post-treatment follow-up are included in Baricitinib 4mg follow up.) | 20 (Participants from treatment who entered the post-treatment follow-up period.)
Completed | 33 | 76 | 20
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Modified Intent-to-Treat (mITT) population: all randomized participants who received at least 1 dose of study drug.
Groups:
- Adalimumab: Adalimumab 40 mg administered by SC injection every 2 weeks through Week 50 and baricitinib placebo orally once daily through Week 52.
  Starting at Week 16, participants who were nonresponders were rescued with baricitinib 4 mg orally once daily through Week 52.
  Participants continued to take background MTX) therapy throughout study.
- Total: Total of all reporting groups
Arm/Group | Placebo | Baricitinib | Adalimumab | Total
Number analyzed (Participants) | 488 | 487 | 330 | 1305
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (11.8) | 53.5 (12.2) | 52.9 (12.3) | 53.3 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 382 | 375 | 251 | 1008
  Male | 106 | 112 | 79 | 297
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 26 | 19 | 18 | 63
  Asian | 148 | 143 | 101 | 392
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 2 | 4 | 10
  White | 302 | 312 | 204 | 818
  More than one race | 7 | 11 | 3 | 21
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 91 | 107 | 57 | 255
  Belgium | 2 | 3 | 3 | 8
  Canada | 5 | 4 | 2 | 11
  China | 21 | 22 | 11 | 54
  Croatia | 1 | 0 | 0 | 1
  Czechia | 16 | 10 | 10 | 36
  France | 8 | 8 | 7 | 23
  Germany | 0 | 0 | 2 | 2
  Greece | 1 | 0 | 2 | 3
  Hungary | 18 | 11 | 8 | 37
  Japan | 93 | 93 | 63 | 249
  South Korea | 21 | 21 | 15 | 57
  Latvia | 2 | 2 | 5 | 9
  Lithuania | 4 | 12 | 10 | 26
  Mexico | 50 | 36 | 39 | 125
  Poland | 26 | 35 | 19 | 80
  Portugal | 1 | 1 | 1 | 3
  Romania | 8 | 6 | 2 | 16
  Russia | 27 | 28 | 23 | 78
  Slovakia | 8 | 8 | 4 | 20
  Slovenia | 4 | 1 | 0 | 5
  South Africa | 24 | 21 | 11 | 56
  Spain | 15 | 11 | 5 | 31
  Taiwan | 6 | 5 | 7 | 18
  United Kingdom | 2 | 6 | 0 | 8
  United States | 34 | 36 | 24 | 94
Duration of Rheumatoid Arthritis [Mean (Standard Deviation); unit: years] | 10.4 (8.7) | 10.3 (8.8) | 9.6 (8.5) | 10.1 (8.7)
Tender Joint Count of 68 Evaluable Joints [Mean (Standard Deviation); unit: Number of Joints] | 23.3 (13.5) | 23.4 (13.0) | 23.4 (13.7) | 23.4 (13.3)
Swollen Joint Count of 66 Evaluable Joints [Mean (Standard Deviation); unit: Number of Joints] | 15.5 (9.4) | 15.0 (8.2) | 15.4 (9.1) | 15.3 (8.9)
High Sensitivity C-Reactive Protein (hsCRP) [Mean (Standard Deviation); unit: milligrams per liter (mg/L)] | 19.66 (20.97) | 22.20 (22.85) | 21.78 (20.83) | 21.14 (21.67)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving American College of Rheumatology 20% Improvement (ACR20)
Description: ACR20 Responder Index is a composite of clinical, laboratory, and functional measures in rheumatoid arthritis (RA). "ACR20 Responder" is a participant who has at least 20% improvement in both tender and swollen joint counts and in at least 3 of the following 5 criteria: Physician's Global Assessment of Disease Activity, Patient's Global Assessment of Disease Activity using visual analog scale (VAS), Health Assessment Questionnaire-Disability Index (HAQ-DI), pain due to arthritis, and high-sensitivity C-reactive protein (hsCRP). Participants with missing responses and participants who discontinued study or drug or were rescued before analysis timepoint were deemed non-responders.
Time Frame: Week 12
Population: Modified Intent-to-Treat (mITT) population: all randomized participants who received at least 1 dose of study drug. Missing values due to discontinuation of study or drug, rescue, or missing data were imputed using nonresponder imputation (NRI).
Measure: Number; unit: percentage of participants
Groups:
- Placebo: Placebo administered orally once daily through Week 24 and placebo administered by SC injection every 2 weeks through Week 50.
  At Week 24, participants were switched to baricitinib 4 mg orally once daily through Week 52.
  Starting at Week 16, participants who were nonresponders were rescued with baricitinib 4 mg orally daily through Week 52.
  Participants continued to take background MTX therapy throughout study.
Arm/Group | Placebo | Baricitinib | Adalimumab
Number analyzed (Participants) | 488 | 487 | 330
percentage of participants | 40.2 | 69.6 | 61.2
Statistical Analysis 1: Comparison: Placebo vs Baricitinib; Test type: Superiority or Other; p = 0.001, Regression, Logistic

2. Secondary Outcome: Change From Baseline in the Modified Total Sharp Score (mTSS)
Description: X-rays of the hands/wrists and feet were scored for structural progression as measured using the mTSS. This methodology quantified the extent of bone erosions and joint space narrowing for 44 and 42 joints, with higher scores representing greater damage.
  The mTSS at a time point is the sum of the erosion (range from 0 to 280) and JSN (range from 0 to 168) scores, for a maximum score of 448.
Time Frame: Baseline, Week 24
Population: mITT population: all randomized participants who received at least 1 dose of study drug and had baseline and at least 1 post-baseline assessments. Missing values due to discontinuation of study, rescue, or missing data were imputed using linear extrapolation (LE).
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Adalimumab: Adalimumab 40 mg administered by SC injection every 2 weeks through Week 50 and baricitinib placebo orally once daily through Week 52.
  Starting at Week 16, participants who are were nonresponders were rescued with baricitinib 4 mg orally once daily through Week 52.
  Participants will continued to take background MTX therapy throughout study.
Arm/Group | Placebo | Baricitinib | Adalimumab
Number analyzed (Participants) | 452 | 470 | 312
units on a scale | 0.84 (2.32) | 0.35 (1.59) | 0.29 (1.47)

3. Secondary Outcome: Change From Baseline in the Health Assessment Questionnaire-Disability Index (HAQ-DI) Score
Description: The HAQ-DI questionnaire assesses the participant's self-perception on the degree of difficulty (0 [without any difficulty], 1 [with some difficulty], 2 [with much difficulty], and 3 [unable to do]) when dressing and grooming, arising, eating, walking, hygiene, reaching, gripping, and performing other daily activities. Scores for each functional area were averaged to calculate the HAQ-DI score, which ranged from 0 (no disability) to 3 (worst disability). A decrease in HAQ-DI score indicated an improvement in the participant's condition.
Time Frame: Baseline, Week 12
Population: mITT population includes all randomized participants who received at least 1 dose of the study drug. Missing values due to discontinuation of study or drug, rescue, or missing data were imputed using modified baseline observation carried forward (mBOCF).
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Baricitinib: Baricitinib 4 mg administered orally once daily through Week 52 and an adalimumab placebo SC injection every 2 weeks through Week 50.
  Starting at Week 16, nonresponder participants originally randomized to baricitinib will continue to receive baricitinib 4 mg administered orally once daily through Week 52.
  Participants will continue to take background MTX therapy throughout study.
- Adalimumab: Adalimumab 40 mg administered by SC injection every 2 weeks through Week 50 and baricitinib placebo orally once daily through Week 52.
  Starting at Week 16, participants who are nonresponders will be rescued with baricitinib 4 mg orally once daily through Week 52.
  Participants will continue to take background MTX therapy throughout study.
Arm/Group | Placebo | Baricitinib | Adalimumab
Number analyzed (Participants) | 488 | 487 | 330
units on a scale | -0.33 (0.51) | -0.65 (0.59) | -0.56 (0.54)

4. Secondary Outcome: Change From Baseline in the Disease Activity Score Based on a 28-Joint Count and High-sensitivity C-reactive Protein (DAS28-hsCRP)
Description: Disease Activity Score (DAS) modified to include 28 joint count (DAS28) consisted of composite score of following variables: tender joint count (TJC28), swollen joint count (SJC28), C-reactive protein (CRP) (milligrams per liter), and Patient's Global Assessment of Disease Activity using visual analog scale (VAS) (participant global VAS). DAS28 was calculated using following formula: DAS28-CRP=0.56*square root (sqrt)(TJC28)+0.28*sqrt(SJC28)+0.36*natural log(CRP+1)+0.014*Patient's Global VAS+0.96. Scores ranged 1.0-9.4, where lower scores indicated less disease activity.
Time Frame: Baseline, Week 12
Population: mITT population includes all randomized participants who received at least 1 dose of the study drug. Missing values due to discontinuation of study or drug, rescue, or missing data were imputed using mBOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Baricitinib: Baricitinib 4 mg administered orally once daily through Week 52 and an adalimumab placebo SC injection every 2 weeks through Week 50.
  Starting at Week 16, nonresponder participants originally randomized to baricitinib continued to receive baricitinib 4 mg administered orally once daily through Week 52.
  Participants continued to take background MTX therapy throughout study.
  .
Arm/Group | Placebo | Baricitinib | Adalimumab
Number analyzed (Participants) | 488 | 487 | 330
units on a scale | -1.01 (1.12) | -2.27 (1.22) | -1.98 (1.28)

5. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 50% (ACR50) and 70% (ACR70) Response
Description: ACR50 and ACR70 Responder Index is a composite of clinical, laboratory, and functional measures in RA. ACR50 and ACR70 Responder is a participant who has at least 50% or 70% improvement, respectively, in both tender and swollen joint counts and in at least 3 of the following 5 criteria: Physician's Global Assessment of Disease Activity, Patient's Global Assessment of Disease Activity, HAQ-DI, pain due to arthritis, and hsCRP.
  Participants with missing responses and participants who discontinued study or drug or were rescued before analysis time point were deemed non-responders.
Time Frame: Week 12, Week 24, Week 52
Population: mITT population: all randomized participants who received at least 1 dose of the study drug. Missing values due to discontinuation of study or drug, rescue, or missing data were imputed using NRI.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Baricitinib | Adalimumab
Number analyzed (Participants) | 488 | 487 | 330
percentage of participants
  ACR50 Week 12 | 16.8 | 45.0 | 34.8
  ACR50 Week 24 | 19.3 | 50.5 | 45.5
  ACR50 Week 52 | NA — No data available. There is no Placebo Arm at week 52. | 55.9 | 47.0
  ACR70 Week 12 | 4.7 | 18.9 | 12.7
  ACR70 Week 24 | 8.0 | 29.8 | 21.8
  ACR70 Week 52 | NA — No data available. There is no Placebo Arm at week 52. | 37.2 | 30.6

6. Secondary Outcome: Change From Baseline in Clinical Disease Activity Index (CDAI) Score
Description: The CDAI is a tool for measurement of disease activity in RA that does not require a laboratory component and was scored by the investigative site. It integrates TJC28 (scored 0-28 with higher scores indicating higher disease activity), SJC28 (scored 0-28 with higher scores indicating higher disease activity), Patient's Global Assessment of Disease Activity (scored on a visual analogue scale from 0-10 cm with higher scores indicating higher disease activity), and Physician's Global Assessment of Disease Activity (scored on a visual analogue scale from 0-10 cm with higher scores indicating higher disease activity). The CDAI is calculated by summing the values of the 4 components. CDAI scores range from 0 to 76; lower scores indicated lower disease activity. A negative change from baseline indicates improvement in condition.
Time Frame: Baseline, Week 12, Week 24, Week 52
Population: mITT population: all randomized participants who received at least 1 dose of the study drug, with a baseline value and at least 1 post-baseline value. Missing values due to discontinuation of study or drug, rescue, or missing data were imputed using modified last observation carried forward (mLOCF).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Baricitinib | Adalimumab
Number analyzed (Participants) | 481 | 478 | 324
units on a scale
  Week 12 | -13.53 (13.88) | -23.00 (12.66) | -20.42 (13.47)
  Week 24 | -14.21 (15.13) | -25.04 (13.61) | -22.92 (14.63)
  Week 52 | NA (NA) — NA= No data available. There is no Placebo Arm at week 52. | -26.44 (14.42) | -23.48 (15.28)

7. Secondary Outcome: Percentage of Participants Achieving Simplified Disease Activity Index (SDAI) Score ≤3.3
Description: SDAI is a tool for measurement of disease activity in RA that integrates TJC28, SJC28, acute phase response using C-reactive protein (milligrams per liter), Patient's Global Assessment of Disease Activity using VAS centimeters (cm), and Physician's Global Assessment of Disease Activity using VAS (cm). The SDAI is calculated by summing the values of the 5 components. Lower scores indicated less disease activity. An index-based definition of remission occurs with an SDAI score ≤3.3.
Time Frame: Week 12, Week 24, Week 52
Population: mITT population: all randomized participants who received at least 1 dose of study drug. Missing values due to discontinuation of study or drug, rescue, or missing data were imputed using NRI.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Baricitinib | Adalimumab
Number analyzed (Participants) | 488 | 487 | 330
percentage of participants
  Week 12 | 1.8 | 8.4 | 7.3
  Week 24 | 3.1 | 16.0 | 13.6
  Week 52 | NA — NA= No data available. There is no Placebo Arm at week 52. | 22.6 | 17.9

8. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology European League Against Rheumatism (ACR/EULAR) Remission - Boolean Remission
Description: The ACR/EULAR definitions of RA remission includes a Boolean-based definition. The Boolean-based definition of remission occurs when all 4 of the following criteria are met at the same visit: TJC28 ≤1, SJC28 ≤1, acute phase response using C-reactive protein (milligrams per deciliter) ≤1, Patient's Global Assessment of Disease Activity using VAS (cm) ≤1.
Time Frame: Week 12, Week 24, Week 52
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Groups:
- Baricitinib: Baricitinib 4 mg administered orally once daily through Week 52 and an adalimumab placebo SC injection every 2 weeks through Week 50.
  Starting at Week 16, nonresponder participants originally randomized to baricitinib continued to receive baricitinib 4 mg administered orally once daily through Week 52.
  Participants continued to take background MTX therapy throughout study.
  Baricitinib: Administered orally
Arm/Group | Placebo | Baricitinib | Adalimumab
Number analyzed (Participants) | 488 | 487 | 330
percentage of participants
  Week 12 | 1.0 | 7.2 | 5.2
  Week 24 | 2.7 | 12.1 | 10.0
  Week 52 | NA — NA= No data available. There is no Placebo Arm at week 52. | 15.6 | 13.0

9. Secondary Outcome: Median of Individual Participant Mean Duration of Morning Joint Stiffness in the Prior 7 Days as Collected in Electronic Diaries
Description: Participants recorded the duration of their morning joint stiffness (MJS) in hours and minutes into electronic diaries daily. If morning joint stiffness duration was longer than 12 hours (720 minutes), it was truncated to 720 minutes for statistical presentations and analyses. The average value across the 7 days preceding each visit was calculated. A decrease in duration of morning joint stiffness indicated an improvement in the participant's condition.
Time Frame: Week 12
Population: mITT population: all randomized participants who received at least 1 dose of the study drug and had at least 4 entries within any post-baseline 7-day window are included in the analysis.
Measure: Median (95% Confidence Interval); unit: Minutes
Arm/Group | Placebo | Baricitinib | Adalimumab
Number analyzed (Participants) | 479 | 479 | 323
Minutes | 60.0 [60.0 to 75.0] | 27.1 [20.0 to 30.0] | 36.6 [30.0 to 45.7]

10. Secondary Outcome: Mean Severity of Morning Joint Stiffness Numeric Rating Scale (NRS) in the Prior 7 Days as Collected in Electronic Diaries
Description: Participants rated the severity of their morning joint stiffness by selecting a number from 0 to 10 that best described their overall level of morning joint stiffness from the time they woke up, where 0 represents "no joint stiffness" and 10 represents "joint stiffness as bad as you can imagine". Participants reported their severity daily in electronic diaries. The average value across the 7 days preceding each visit was calculated.
Time Frame: Week 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Baricitinib | Adalimumab
Number analyzed (Participants) | 479 | 479 | 323
units on a scale | 4.1 (2.3) | 3.0 (2.2) | 3.4 (2.3)

11. Secondary Outcome: Mean Worst Tiredness Numeric Rating Scale (NRS) in the Prior 7 Days as Collected in Electronic Diaries
Description: Participants rated their tiredness by selecting a number from 0 to 10 that best described their worst tiredness during the last 24 hours, where 0 represents "no tiredness" and 10 represents "as bad as you can imagine". Participants reported their worst tiredness in electronic diaries. The average value across the 7 days preceding each visit is calculated.
Time Frame: Week 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Baricitinib | Adalimumab
Number analyzed (Participants) | 479 | 479 | 323
units on a scale | 4.4 (2.3) | 3.6 (2.2) | 3.9 (2.3)

12. Secondary Outcome: Mean Worst Joint Pain NRS in the Prior 7 Days as Collected in Electronic Diaries
Description: Participants rated their joint pain by selecting a number from 0 to 10 that best described their worst joint pain during the last 24 hours, where 0 represents "no pain" and 10 represents "pain as bad as you can imagine". Participants reported their worst joint pain in daily electronic diaries. The average value across the 7 days preceding each visit was calculated.
Time Frame: Week 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Baricitinib | Adalimumab
Number analyzed (Participants) | 479 | 479 | 323
units on a scale | 4.6 (2.2) | 3.4 (2.2) | 4.0 (2.3)

13. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Scale Scores
Description: The Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Scale is a brief 13-item, symptom-specific questionnaire that specifically assesses the participant's self-reported severity of fatigue and its impact upon daily activities and functioning. The FACIT-F uses a numeric rating scale of 0 ("Not at all") to 4 ("Very much") for each item to assess fatigue and its impact in the past 7 days. Total scores range from 0 to 52, with higher scores indicating less fatigue.
Time Frame: Baseline, Week 12, Week 24, Week 52
Population: mITT population: all randomized participants who received at least 1 dose of study drug, with a baseline value and at least 1 post-baseline value. Missing values due to discontinuation of study or drug, rescue, or missing data were imputed using mLOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Baricitinib | Adalimumab
Number analyzed (Participants) | 475 | 479 | 320
units on a scale
  Week 12 | 6.8 (9.9) | 9.6 (10.4) | 9.5 (10.1)
  Week 24 | 6.6 (10.4) | 10.4 (10.8) | 9.9 (11.2)
  Week 52 | NA (NA) — NA= No data available. There is no Placebo Arm at week 52. | 10.8 (10.9) | 9.8 (10.8)

14. Secondary Outcome: Change From Baseline in Mental Component Score (MCS), Physical Component Score (PCS) of the Medical Outcomes Study 36-Item Short Form Health Survey Version 2 Acute (SF-36v2 Acute)
Description: The SF-36 is a health-related survey that assesses participant's quality of life and consists of 36 questions covering 8 health domains: physical functioning, bodily pain, role limitations due to physical problems and emotional problems, general health, mental health, social functioning, vitality, and 2 component scores (mental [MCS] and physical [PCS]). MCS consisted of social functioning, vitality, mental health, and role-emotional scales. PCS consisted of physical functioning, bodily pain, role-physical, and general health scales. Each domain is scored by summing the individual items and transforming the scores into a 0 to 100 scale with higher scores indicating better health status or functioning.
Time Frame: Baseline, Week 12, Week 24, Week 52
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Baricitinib | Adalimumab
Number analyzed (Participants) | 475 | 479 | 320
units on a scale
  MCS Week 12 | 3.2 (10.3) | 3.3 (10.5) | 3.8 (10.8)
  MCS Week 24 | 2.2 (11.4) | 3.8 (10.9) | 3.9 (11.6)
  MCS Week 52 | NA (NA) — No data available. There is no Placebo Arm at week 52. | 4.0 (10.8) | 3.7 (11.2)
  PCS Week 12 | 4.3 (7.1) | 8.9 (8.1) | 7.6 (8.2)
  PCS Week 24 | 4.6 (7.8) | 9.9 (8.2) | 8.3 (9.1)
  PCS Week 52 | NA (NA) — No data available. There is no Placebo Arm at week 52. | 10.4 (9.0) | 9.0 (9.2)

15. Secondary Outcome: Change From Baseline in European Quality of Life-5 Dimensions-5 Level (EQ-5D-5L) Scores
Description: European Quality of Life-5 Dimensions-5 Level (EQ-5D-5L) is a standardized measure of health status of the participant. One component consists of a descriptive system of the respondent's health comprised of the following 5 participant-reported dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The responses are used to derive the health state index scores using the United Kingdom (UK) algorithm, with scores ranging from -0.594 to 1, and the United States (US) algorithm, with scores ranging from -0.109 to 1. A higher score indicates better health state.
Time Frame: Baseline, Week 12, Week 24, Week 52
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Baricitinib | Adalimumab
Number analyzed (Participants) | 475 | 479 | 320
units on a scale
  Index Score (US Algorithm) Week 12 | 0.073 (0.151) | 0.132 (0.156) | 0.130 (0.159)
  Index Score (US Algorithm) Week 24 | 0.065 (0.168) | 0.143 (0.168) | 0.137 (0.167)
  Index Score (US Algorithm) Week 52 | NA (NA) — NA= No data available. There is no Placebo Arm at week 52. | 0.152 (0.163) | 0.141 (0.189)
  Index Score (UK Algorithm) Week 12 | 0.107 (0.221) | 0.188 (0.228) | 0.186 (0.232)
  Index Score (UK Algorithm) Week 24 | 0.094 (0.247) | 0.203 (0.244) | 0.195 (0.245)
  Index Score (UK Algorithm) Week 52 | NA (NA) — NA= No data available. There is no Placebo Arm at week 52. | 0.215 (0.235) | 0.198 (0.273)

16. Secondary Outcome: Change From Baseline in European Quality of Life-5 Dimensions-5 Level (EQ-5D-5L) Scores (Self-Perceived Health)
Description: A second component of the EQ-5D-5L is a self-perceived health score which is assessed using a VAS that ranges from 0 to 100 millimeter (mm), where 0 indicates the worst health you can imagine and 100 indicates the best health you can imagine.
Time Frame: Baseline, Week 12, Week 24, Week 52
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Placebo | Baricitinib | Adalimumab
Number analyzed (Participants) | 475 | 479 | 320
millimeter
  Self-Perceived Health Week 12 | 7.9 (26.2) | 14.9 (25.8) | 10.7 (26.9)
  Self-Perceived Health Week 24 | 5.6 (27.1) | 17.5 (28.3) | 12.6 (28.9)
  Self-Perceived Health Week 52 | NA (NA) — NA= No data available. There is no Placebo Arm at week 52. | 19.9 (28.0) | 13.3 (29.7)

17. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment-Rheumatoid Arthritis (WPAI-RA) Scores
Description: The Work Productivity and Activity Impairment-Rheumatoid Arthritis (WPAI-RA) questionnaire was developed to measure the effect of general health and symptom severity on work productivity and regular activities in the 7 days prior to the visit. It contains 6 items covering overall work productivity (health), overall work productivity (symptom), impairment of regular activities (health), and impairment of regular activities (symptom). Scores are calculated as impairment percentages. The WPAI-RA yields four types of scores: Absenteeism (work time missed), Presenteeism (impairment at work), Work productivity loss (overall work impairment), and Activity impairment.
Time Frame: Baseline, Week 12, Week 24, Week 52
Population: mITT population includes all randomized participants who received at least 1 dose of the study drug, with a baseline value and an observed value at the time point being summarized.
Measure: Mean (Standard Deviation); unit: percentage of impairment
Arm/Group | Placebo | Baricitinib | Adalimumab
Number analyzed (Participants) | 458 | 474 | 315
percentage of impairment
  Absenteeism Week 12 (n=160,168,118) | 0.5 (27.7) | -4.9 (20.6) | -0.5 (25.7)
  Absenteeism Week 24 (n=118,139,102) | -1.6 (24.5) | -1.8 (25.2) | -3.2 (23.8)
  Absenteeism Week 52 (n=0,124,92) | NA (NA) — NA= No data available. There is no Placebo Arm at week 52. | -3.8 (25.1) | -3.7 (24.3)
  Presenteeism Week 12 (n=147,160,113) | -11 (23) | -21 (26) | -16 (24)
  Presenteeism Week 24 (n=110,134,99) | -11 (22) | -23 (27) | -22 (26)
  Presenteeism Week 52 (n=0,119,88) | NA (NA) — NA= No data available. There is no Placebo Arm at week 52. | -25 (27) | -25 (27)
  Work Productivity Loss Week 12 (n=147,160,113) | -10.4 (24.3) | -21.6 (28.0) | -14.0 (25.6)
  Work Productivity Loss Week 24 (n=110,134,99) | -9.0 (24.9) | -22.1 (30.2) | -21.4 (27.2)
  Work Productivity Loss Week 52 (n=0,119,88) | NA (NA) — NA= No data available. There is no Placebo Arm at week 52. | -24.4 (30.1) | -24.6 (29.8)
  Activity Impairment Week 12 (n=458,474,315) | -11 (25) | -25 (26) | -20 (25)
  Activity Impairment Week 24 (n=333,430,272) | -16 (26) | -28 (27) | -26 (26)
  Activity Impairment Week 52 (n=0,396,240) | NA (NA) — NA= No data available. There is no Placebo Arm at week 52. | -30 (27) | -28 (27)

18. Secondary Outcome: Change From Baseline in Joint Space Narrowing (JSN) and Bone Erosion Scores
Description: X-rays of the hands/wrists and feet were assessed for joint space narrowing (JSN) and bone erosions. Assessment of JSN for each hand (15 joints per hand) and foot (6 joints per foot), including subluxation, is scored from 0 to 4, with 0 indicating no (normal) JSN and 4 indicating complete loss of joint space, bony ankylosis or luxation. JSN scores ranged from 0-168. A score of 0 would indicate no change and higher scores represent a worsening of joint space narrowing.
  The bone erosion score is a summary of erosion severity in 32 joints of the hands and 12 joints of the feet. Each joint is scored according to the surface area involved from 0 to 5 for hand joints and 0 to 10 for the foot joints, with 0 indicating no erosion and the highest score (5 for the hand and 10 for the foot) indicating extensive loss of bone from more than one half of the articulating bone. Erosion scores ranged from 0 (no erosion) to 280 (high erosion).
Time Frame: Baseline, Week 24, Week 52
Population: mITT population: all randomized participants who received at least 1 dose of study drug and had baseline and at least 1 post-baseline assessment. Missing values due to discontinuation of study, rescue, or missing data were imputed using LE.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Baricitinib | Adalimumab
Number analyzed (Participants) | 452 | 473 | 312
units on a scale
  Joint Space Narrowing Week 24 (n= 452, 470, 312) | 0.27 (1.15) | 0.10 (0.74) | 0.09 (0.52)
  Joint Space Narrowing Week 52 (n= 452, 473, 312) | 0.56 (2.33) | 0.18 (1.02) | 0.17 (1.00)
  Bone Erosion Score Week 24 (n=452, 470, 312) | 0.57 (1.58) | 0.25 (1.12) | 0.20 (1.08)
  Bone Erosion Score Week 52 (n= 452, 473, 312) | 1.15 (3.21) | 0.42 (1.91) | 0.34 (2.00)

19. Secondary Outcome: Population Pharmacokinetics (PK): Peak Concentration at Steady State (Cmax,ss) of Baricitinib
Time Frame: Week 0: 15 and 60 minutes postdose; Week 4: 2 to 4 hours post-dose; Week 8: 4 to 6 hours post-dose; Week 12; Week 12; Week 24; Week 32: Pre-dose
Population: All randomized participants who received at least 1 dose of study drug (during study or rescue treatment) with evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole/Liter (nmol/L)
Groups:
- Baricitinib: Baricitinib 4 mg administered orally once daily through Week 52
Arm/Group | Baricitinib
Number analyzed (Participants) | 635
nanomole/Liter (nmol/L) | 143 (19.7)

20. Secondary Outcome: Population PK: Area Under the Concentration Versus Time Curve at a Dosing Interval at Steady State (AUCtau,ss) of Baricitinib
Time Frame: as for outcome 19
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole*hr/Liter (nmol*hr/L)
Arm/Group | Baricitinib
Number analyzed (Participants) | 635
nanomole*hr/Liter (nmol*hr/L) | 1220 (45.8)

ADVERSE EVENTS:
Description: All enrolled participants including rescue therapy. After Week 16, rescue therapy will be offered at the discretion of the investigator based on tender joint count and swollen joint count.
Groups:
- Placebo Treatment A: Placebo Treatment A (week 0-24).
  Placebo administered orally (PO) once daily (QD) through Week 24 and placebo administered by subcutaneous (SC) injection every 2 weeks through Week 50.
  At Week 24, participants were given baricitinib 4 milligram (mg) orally once daily through Week 52.
  Starting at Week 16, participants who were nonresponders were rescued with baricitinib 4 mg orally once daily through Week 52.
- Baricitinib Treatment A: Baricitinib Treatment A (week 0-24).
  Baricitinib 4 mg administered orally once daily through Week 52 and an adalimumab placebo SC injection every 2 weeks through Week 50.
  Starting at Week 16, nonresponder participants originally randomized to baricitinib continued to receive baricitinib 4 mg administered orally once daily through Week 52.
- Adalimumab Treatment A: Adalimumab Treatment A (week 0-24).
  Adalimumab 40 mg administered by SC injection every 2 weeks through Week 50 and baricitinib placebo orally once daily through Week 52.
  Starting at Week 16, participants who were nonresponders were rescued with baricitinib 4 mg orally once daily through Week 52.
- Placebo Treatment B: Placebo Treatment B (week 24-52).
  Placebo administered orally (PO) once daily (QD) through Week 24 and placebo administered by subcutaneous (SC) injection every 2 weeks through Week 50.
  At Week 24, participants were given baricitinib 4 milligram (mg) orally once daily through Week 52.
  Starting at Week 16, participants who were nonresponders were rescued with baricitinib 4 mg orally once daily through Week 52.
- BaricitinibTreatment B: Baricitinib Treatment B (week 24-52).
  Baricitinib 4 mg administered orally once daily through Week 52 and an adalimumab placebo SC injection every 2 weeks through Week 50.
  Starting at Week 16, nonresponder participants originally randomized to baricitinib continued to receive baricitinib 4 mg administered orally once daily through Week 52.
- Adalimumab Treatment B: Adalimumab Treatment B (week 24-52).
  Adalimumab 40 mg administered by SC injection every 2 weeks through Week 50 and baricitinib placebo orally once daily through Week 52.
  Starting at Week 16, participants who were nonresponders were rescued with baricitinib 4 mg orally once daily through Week 52.
- Rescue: Baricitinib 4 mg administered PO QD through Week 52 (Week 16-52).
- Placebo Follow-up; Adalimumab Follow-up: No study drug received. Participants return for safety follow-up visit 28 days after the last dose of study drug.
- Baricitinib Follow-up: No study drug received. Participants return for safety follow-up visit 28 days after the last dose of study drug. Participants who were rescued or switched to Baricitinib 4 mg.
Arm/Group | Placebo Treatment A | Baricitinib Treatment A | Adalimumab Treatment A | Placebo Treatment B | BaricitinibTreatment B | Adalimumab Treatment B | Rescue | Placebo Follow-up | Baricitinib Follow-up | Adalimumab Follow-up
Serious Adverse Events (participants affected / at risk) | 26/488 | 26/487 | 7/330 | 12/306 | 16/424 | 9/267 | 17/227 | 2/33 | 0/76 | 0/20
Other Adverse Events (participants affected / at risk) | 177/488 | 196/487 | 132/330 | 58/306 | 70/424 | 38/267 | 46/227 | 3/33 | 0/76 | 3/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Treatment A (N=488) | Baricitinib Treatment A (N=487) | Adalimumab Treatment A (N=330) | Placebo Treatment B (N=306) | BaricitinibTreatment B (N=424) | Adalimumab Treatment B (N=267) | Rescue (N=227) | Placebo Follow-up (N=33) | Baricitinib Follow-up (N=76) | Adalimumab Follow-up (N=20)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Lymphocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Macular fibrosis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jejunal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangitis sclerosing (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis infective (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disseminated tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epiglottitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atypical pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia pseudomonal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post concussion syndrome (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung squamous cell carcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalised anxiety disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrosclerosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal septum perforation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hysterectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fracture treatment (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo Treatment A (N=488) | Baricitinib Treatment A (N=487) | Adalimumab Treatment A (N=330) | Placebo Treatment B (N=306) | BaricitinibTreatment B (N=424) | Adalimumab Treatment B (N=267) | Rescue (N=227) | Placebo Follow-up (N=33) | Baricitinib Follow-up (N=76) | Adalimumab Follow-up (N=20)
Anaemia (Blood and lymphatic system disorders) | 15 (16) | 16 (16) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 8 (9) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 14 (16) | 11 (12) | 8 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 7 (7) | 9 (9) | 8 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (7) | 14 (15) | 9 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 14 (14) | 19 (22) | 8 (8) | 11 (12) | 12 (12) | 5 (5) | 6 (7) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 4 (5) | 12 (12) | 5 (5) | 3 (3) | 10 (10) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 35 (39) | 37 (41) | 34 (40) | 15 (19) | 24 (26) | 14 (15) | 9 (11) | 2 (2) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 14 (14) | 12 (13) | 12 (12) | 10 (12) | 4 (4) | 7 (7) | 5 (10) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 14 (15) | 15 (17) | 13 (16) | 10 (10) | 13 (13) | 4 (4) | 6 (7) | 0 (0) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 16 (16) | 21 (25) | 13 (14) | 5 (5) | 10 (10) | 5 (6) | 5 (6) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 5 (5) | 8 (9) | 9 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 3 (3) | 13 (15) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 7 (7) | 15 (15) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 (2) | 10 (11) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 9 (9) | 10 (13) | 7 (7) | 9 (9) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 14 (15) | 5 (6) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 12 (12) | 14 (17) | 13 (16) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2/79 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 7 (7) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 5 (6) | 3 (3) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 13 (13) | 9 (9) | 11 (11) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 1 (1) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1/47 (1) | 0 (0) | 0 (0) | 0 (0)
Calculus prostatic (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1/47 (1) | 0 (0) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 1 (1) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1/16 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days